CLINICAL TRIAL: NCT00813319
Title: Overcoming Barriers to Vaccination With GARDASIL in Underserved Girls and Adolescents
Brief Title: Girls OnGuard: HPV Vaccination Uptake Among African American Adolescent Females
Acronym: Girls OnGuard
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00015576; Merck - Emory UPN 08042902 (Other: Other)
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2014-08-12 (Estimated); Status verified 2014-08

CONDITIONS: Vaccination
Keywords: GARDASIL; HPV; Vaccination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Girls OnGuard/HPV awareness (Experimental): Adolescents will watch a short (10 min), interactive DVD designed to promote HPV awareness and initial GARDASIL vaccination and receive a keepsake to help them remember to return to the clinic for their second and third vaccine doses.
  Interventions: Behavioral: Girls OnGuard
- 2 - General health promotion (No Intervention): Adolescents will watch an equally short (10 min) DVD on healthy lifestyles and behaviors. HPV awareness and vaccination will not be addressed.

INTERVENTIONS:
Behavioral: Girls OnGuard — Using the Information-Motivation-Behavioral Skills Model (IMB) as a framework, Girls OnGuard is an interactive,culturally-appropriate, computer-delivered program design to enhance initial uptake of GARDASIL by addressing three major components: (1) information about GARDASIL; (2) motivation to obtain GARDASIL vaccination; and (3) behavioral skills to enhance self-efficacy of obtaining GARDASIL vaccination.
  Arms: 1 - Girls OnGuard/HPV awareness

SUMMARY:
African American adolescent females seeking treatment for STIs are an underserved population at increased risk for HPV infection. While GARDASIL is an effective preventive vaccine, vaccination rates are low. Given the risk for HPV infection among this subgroup and the negative health effects associated with HPV, enhancing uptake of GARDASIL is necessary. The goal of this project is to promote GARDASIL vaccination through the development of a new multi-component, culturally-appropriate, interactive DVD.

We propose to recruit 280 unmarried African American adolescent females, 13-18 years of age, from participating clinic sites in Atlanta, Georgia. While seeking clinical services, adolescents will be contacted and invited to participate in the proposed study. Eligible adolescents will be required to provide written assent/consent prior to participation. Adolescents who are eligible and willing to participate in the project will complete a short survey on a laptop computer. The survey is designed to assess adolescents' risk taking and preventive behaviors. After they complete the survey, adolescents will be assigned at random to one of two groups. In one group, adolescents will watch a short (10 min), interactive DVD designed to promote HPV awareness and initial GARDASIL vaccination and receive a keepsake to help them remember to return to the clinic for their second and third vaccine doses. In the second group, adolescents will watch an equally short (10 min) DVD on healthy lifestyles and behaviors. All adolescents are eligible to receive the GARDASIL vaccine at participating study clinics as part of their routine standard of care.

With the help of clinic staff, participant medical records will be reviewed over a 7 month period to assess vaccination rates. Vaccination rates from adolescents who received the interactive HPV/GARDASIL awareness DVD will be compared to the group of adolescents who received the healthy lifestyles DVD. It is hypothesized that study participants receiving the interactive DVD intervention that promotes HPV awareness will have higher vaccination rates over time.

ELIGIBILITY:
Inclusion Criteria:

* African American
* Female
* Age 13-18 years
* Seeking reproductive/STI services at participating clinic
* Ability to give written informed consent or assent

Exclusion Criteria:

* Pregnant
* Married
* Already received the HPV vaccine

Ages: 13 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J. DiClemente, PhD, Principal Investigator — Emory University Rollins School of Public Health
Locations (2):
- United States (2):
  - Fulton County Department of Health and Wellness, Atlanta, Georgia
  - DeKalb County Health Department, Decatur, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion
Started | 108 | 108
Completed | 108 (100 out of 108 have complete follow-up data, there were 8 missing charts 7 months post-randomization) | 108 (104 out of 108 have complete follow-up data, there were 4 missing charts 7 months post-randomization)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion | Total
Number analyzed (Participants) | 108 | 108 | 216
Age, Continuous [Mean (Standard Deviation); unit: Years] | 16.68 (1.44) | 16.26 (1.54) | 16.47 (1.50)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 108 | 108 | 216
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 108 | 216
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 108 | 108 | 216

OUTCOME MEASURES:

1. Primary Outcome: GARDASIL Vaccination Uptake and Compliance With Second and Third Doses
Description: Number of participants who received at least 1 dose, 2 doses, 3 doses
Time Frame: measured at 7 months post-randomization
Measure: Number; unit: participants
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion
Number analyzed (Participants) | 100 | 104
participants
  Number of participants who received at least 1 dos | 12 | 12
  Number of participants who received 2 doses | 8 | 3
  Number of participants who received 3 doses | 6 | 2
Statistical Analysis 1: Comparison: 1 - Girls OnGuard/HPV Awareness vs 2 - General Health Promotion; This comparison is for participants in the Girls OnGuard/HPV Awareness condition compared to the General Health Promotion condition; Test type: Superiority or Other; p > .05, Chi-squared

2. Secondary Outcome: STD Incidence
Description: Number of participants who tested positive for any STD 7 months post randomization, information was gathered via medical chart abstraction
Time Frame: 7 months post randomization
Measure: Number; unit: participants
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion
Number analyzed (Participants) | 100 | 104
participants | 35 | 32
Statistical Analysis 1: Comparison: 1 - Girls OnGuard/HPV Awareness vs 2 - General Health Promotion; Test type: Superiority or Other; p = .52, Chi-squared

3. Primary Outcome: Total Doses Received of HPV Vaccine
Description: As an additional primary outcome, we assessed the total number of vaccine doses received
Time Frame: measured at 7-months post randomization
Measure: Number; unit: Doses
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion
Number analyzed (Participants) | 100 | 104
Doses | 26 | 17
Statistical Analysis 1: Comparison: 1 - Girls OnGuard/HPV Awareness vs 2 - General Health Promotion; This comparison is for total doses received (26 in Girls OnGuard/HPV Awareness condition compared to 17 in General Health Promotion condition); Test type: Superiority or Other; p = .12, Chi-squared; Degrees of freedom = 2

ADVERSE EVENTS:
Arm/Group | 1 - Girls OnGuard/HPV Awareness | 2 - General Health Promotion
Serious Adverse Events (participants affected / at risk) | 0/108 | 0/108
Other Adverse Events (participants affected / at risk) | 0/108 | 0/108

LIMITATIONS AND CAVEATS:
Limited sample size; Brevity of the computer-administered intervention; Substantial variability between and within clinics with respect to patient-provider interactions; Lack of a follow-up assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No